CLINICAL TRIAL: NCT03152019
Title: Efficacy and Safety of a 0.1% Tacrolimus Nasal Ointment as a Treatment for Epistaxis in Hemorrhagic Hereditary Telangiectasia (HHT) - A Double Blind, Randomized, Placebo-controlled, Multicenter Trial
Brief Title: Efficacy and Safety of a 0.1% Tacrolimus Nasal Ointment as a Treatment for Epistaxis in Hemorrhagic Hereditary Telangiectasia (HHT)
Acronym: TACRO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 69HCL16_0705; 2017-000085-30 (EudraCT Number)
Record Dates: First submitted 2017-05-11; First posted 2017-05-12 (Actual); Results first posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2019-07

CONDITIONS: Hemorrhagic Hereditary Telangiectasia (HHT)
Keywords: Hemorrhagic Hereditary Telangiectasia (HHT); Antiangiogenic therapy; Tacrolimus
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — Tacrolimus; Ointments

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protopic® 0.1% (Tacrolimus) ointment (Active Comparator): Protopic® 0.1% ointment, packed in blinded tube of 30g.
  Interventions: Drug: Protopic® (Tacrolimus) 0.1% ointment
- Placebo ointment (Placebo Comparator): Same formulation as the Protopic® 0.1% ointment but without tacrolimus, packed in blinded tube of 30g.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Protopic® (Tacrolimus) 0.1% ointment — About 0,1g of ointment is administered by the patient on nasal mucosa of each nostril twice a day for 6 weeks.
  Arms: Protopic® 0.1% (Tacrolimus) ointment
Drug: Placebo — About 0,1g of ointment is administered by the patient on nasal mucosa of each nostril twice a day for 6 weeks.
  Arms: Placebo ointment

SUMMARY:
The recognized manifestations of HHT are all due to abnormalities in vascular structure. Epistaxis due to telangiectases formation is spontaneous, very variable, recurrent in 90% of patients, and associated with severe anemia in 2-10%. They also significantly reduce quality of life.

Improvement in epistaxis has been shown in HHT patients after a liver transplantation. It was hypothesized that the immunosuppressive treatment (FK506) used to prevent rejection may have an anti-angiogenic effect.

The results of Albiñana et al suggest that the mechanism of action of FK506 involves a partial correction of endoglin and ALK1 haplosufficiency, genes responsible for 90% of HHT case.

Tacrolimus ointment is available on the market for the treatment of eczema and can therefore readily be used as it is for nasal administration. Topical nasal administration of tacrolimus may be an easy local ENT treatment that is non-aggressive and results in little trauma for the patient in relation to other first line treatment possibilities.

The main objective of this trial is to evaluate, at 6 weeks after the end of the treatment, the efficacy on the duration of nosebleeds, of 6 weeks tacrolimus nasal ointment application, in patients with HHT complicated by nosebleeds (30 min/6 weeks). Secondary objectives are to evaluate the tolerance throughout the study, the efficacy on anemia and on clinical parameters (nosebleeds, quality of life, epistaxis severity score questionnaire and blood transfusions) and the systemic absorption of nasal administration.

This is a multicenter prospective and double blinded phase I/II trial. A total of 48 patients will be randomized versus placebo using an allocation ratio of 1:1. The ointment (Protopic® at 0.1% or placebo) will be self-administered by the patient with one administration in each nostril twice a day for 6 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients who have given their free, informed and signed consent.
* Patients affiliated to a social security scheme or similar.
* Patients monitored for clinically confirmed HHT (presence of at least 3 Curaçao criteria) and/or confirmed by molecular biology.
* Patient presenting nosebleeds with total duration > 30 minutes for 6 weeks prior to the time of inclusion justified by completed follow-up grids.

Exclusion Criteria:

* Women who are pregnant or nursing (lactating), women of child-bearing potential without reliable contraception.
* Patients not affiliated to a social security scheme.
* Patients who are protected adults under the terms of the law (French Public Health Code).
* Refusal to consent.
* Patients for whom the diagnosis of HHT has not been confirmed clinically and/or by molecular biology.
* Participation in another clinical trial which may interfere with the proposed trial (judgment of the investigator).
* Patients who have undergone nasal surgery in the 6 weeks prior to inclusion.
* Known hypersensitivity to macrolides in general, to tacrolimus or to any of the excipients.
* Patient with an inherited skin barrier disease such as Netherton's syndrome, lamellar ichtyosis, generalized erythroderma, graft-versus-host skin disease, or suffering from generalized erythroderma.
* Patient with CYP3A4 inhibitors treatment, e.g. erythromycin, itraconazole, ketoconazole and diltiazem.
* Patients who have incompletely filled in the nosebleed grids in the 10 weeks preceding the treatment. If there is missing data for more than 7 days, the patient cannot be included.
* Patients who do not present nosebleeds with a total duration of > 30 minutes for 6 weeks prior to the time of inclusion.
* Patients with ongoing immunosuppressive treatment.
* Patients with known and symptomatic immune deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie DUPUIS-GIROD, Principal Investigator — Hospices Civils de Lyon Centre de Référence pour la maladie de Rendu-Osler Service de génétique Clinique Bâtiment A1 - HFME; Sophie DUPUIS-GIROD, Principal Investigator — Hospices Civils de Lyon
Locations (3):
- France (3):
  - Hôpital Femme Mère Enfant, Bron
  - CHU Estaing, Clermont-Ferrand
  - CHU de Montpellier, Montpellier

REFERENCES:
- See also: Related Info — http://www.rendu-osler.fr

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Protopic® 0.1% (Tacrolimus) Ointment | Placebo Ointment
Started | 25 | 25
Completed | 25 | 24
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: n=26 included in per protocol analysis because of a wrong allocation: 1 patient in placebo group who received tacrolimus
Groups:
- Total: Total of all reporting groups
Arm/Group | Protopic® 0.1% (Tacrolimus) Ointment | Placebo Ointment | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 23 | 49
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 17 | 10 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 26 | 24 | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Experiencing an Improvement in Their Nosebleeds
Description: Efficacy of tacrolimus nasal ointment on nosebleeds when administered for 6 weeks
Time Frame: up to 12 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Protopic® 0.1% (Tacrolimus) Ointment | Placebo Ointment
Number analyzed (Participants) | 26 | 24
Participants | 10 | 9
Statistical Analysis 1: Comparison: Protopic® 0.1% (Tacrolimus) Ointment vs Placebo Ointment; Test type: Superiority; p < 0.05, Chi-squared; percentages = 0.77

2. Secondary Outcome: Adverse Events
Description: Tolerance will be evaluated by recording adverse reactions and adverse events during the treatment period and the follow up period and by clinical examinations during the follow-up period.
Time Frame: up to 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Number of Epistaxis
Description: Evaluate efficacy on clinical criteria : epistaxis frequency before and after treatment.
Time Frame: up to 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Epistaxis Duration
Description: To evaluate efficacy of tacrolimus nasal ointment on duration of nosebleeds before and after treatment.
Time Frame: up to 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Hemoglobin Level
Description: before and after treatment.
Time Frame: up to 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Ferritin Level
Description: before and after treatment.
Time Frame: up to 12 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Quality of Life Assessed by SF36 Questionnaire
Description: To evaluate efficacy on quality of life with SF36 before and after treatment
Time Frame: up to 12 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Severity Epistaxis Score Assessed by ESS Questionnaire
Description: To evaluate efficacy on severity epistaxis score with ESS before and after treatment.
Time Frame: up to 12 weeks
Reporting Status: Not Posted

9. Secondary Outcome: The Percentage of Patient With Tacrolimus Detection in the Blood
Description: To evaluate systemic absorption after tacrolimus nasal administrations.
Time Frame: up to 6 weeks
Reporting Status: Not Posted

10. Secondary Outcome: the Level of Exposure of Patient With Tacrolimus Detection in the Blood.
Description: To evaluate systemic absorption after tacrolimus nasal administrations.
Time Frame: up to 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Day 0, day 15, day 31, day 43, day 85
Description: n=26 in PP because of a wrong allocation, 1 patient in placebo group who received tacrolimus
Arm/Group | Protopic® 0.1% (Tacrolimus) Ointment | Placebo Ointment
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/26 | 2/24
Other Adverse Events (participants affected / at risk) | 11/26 | 8/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Protopic® 0.1% (Tacrolimus) Ointment (N=26) | Placebo Ointment (N=24)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Protopic® 0.1% (Tacrolimus) Ointment (N=26) | Placebo Ointment (N=24)
Thermal burn (Injury, poisoning and procedural complications) | 9 (10) | 3 (3)
parosmia (Nervous system disorders) | 2 (2) | 0 (0)
malaise (General disorders) | 0 (0) | 3 (3)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/19/NCT03152019/Prot_SAP_000.pdf